CLINICAL TRIAL: NCT03083457
Title: Physiological Effects of Positive End-expiratory Pressure With or Without Recruiting Maneuvers in Patients Receiving Low-tidal Volume Ventilation During General Anesthesia for Open Abdominal Surgery. A Randomized, Cross-over Study
Brief Title: Physiological Effects of Lung Recruitment During General Anesthesia and Low-tidal Volume Ventilation
Acronym: PEEP-RM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Massimo Antonelli, MD, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 10989/15
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia, General; Surgery
MeSH Terms: interventions — Anesthetics, General; Hypodermoclysis

STUDY DESIGN:
Intervention Model Description: Each patient will be randomized to receive or not scheduled recruiting maneuvers every hour. In each of the two groups, patients will receive mechanical ventilation with 3 different levels of PEEP in a sequential, randomized, cross-over manner: each period will last 40 minutes.
  A randomization sequence will be produced by a dedicated software and sealed envelopes will be used to allocate patients to study treatments.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PEEP2 + RM (Experimental): General anesthetic, 40 minutes of Low-tidal volume ventilation with PEEP=2 cmH2O and scheduled recruiting maneuvers at the beginning of each PEEP step, continuous fluid administration at a standard dose, fluid resuscitation or amine administration if deemed necessary by the attending physician blinded to the design of the study
  Interventions: Drug: Fluid resuscitation or amine administration; Drug: General anesthetic; Drug: Fluid administration; Procedure: Low-tidal volume ventilation; Procedure: Scheduled recruiting maneuvers
- PEEP7 + RM (Experimental): General anesthetic, 40 minutes of Low-tidal volume ventilation with PEEP=7 cmH2O and scheduled recruiting maneuvers at the beginning of the PEEP step, continuous fluid administration at a standard dose, fluid resuscitation or amine administration if deemed necessary by the attending physician blinded to the design of the study
  Interventions: Drug: Fluid resuscitation or amine administration; Drug: General anesthetic; Drug: Fluid administration; Procedure: Low-tidal volume ventilation; Procedure: Scheduled recruiting maneuvers
- PEEP12 + RM (Experimental): General anesthetic, 40 minutes of Low-tidal volume ventilation with PEEP=12 cmH2O and scheduled recruiting maneuvers at the beginning of the PEEP step, continuous fluid administration at a standard dose, fluid resuscitation or amine administration if deemed necessary by the attending physician blinded to the design of the study
  Interventions: Drug: Fluid resuscitation or amine administration; Drug: General anesthetic; Drug: Fluid administration; Procedure: Low-tidal volume ventilation; Procedure: Scheduled recruiting maneuvers
- PEEP2 - RM (Experimental): General anesthetic, 40 minutes of Low-tidal volume ventilation with PEEP=2 cmH2O, continuous fluid administration at a standard dose, fluid resuscitation or amine administration if deemed necessary by the attending physician blinded to the design of the study
  Interventions: Drug: Fluid resuscitation or amine administration; Drug: General anesthetic; Drug: Fluid administration; Procedure: Low-tidal volume ventilation
- PEEP7 - RM (Experimental): General anesthetic, 40 minutes of Low-tidal volume ventilation with PEEP=7 cmH2O, continuous fluid administration at a standard dose, fluid resuscitation or amine administration if deemed necessary by the attending physician blinded to the design of the study
  Interventions: Drug: Fluid resuscitation or amine administration; Drug: General anesthetic; Drug: Fluid administration; Procedure: Low-tidal volume ventilation
- PEEP12 - RM. (Experimental): General anesthetic, 40 minutes of Low-tidal volume ventilation with PEEP=12 cmH2O, continuous fluid administration at a standard dose, fluid resuscitation or amine administration if deemed necessary by the attending physician blinded to the design of the study
  Interventions: Drug: Fluid resuscitation or amine administration; Drug: General anesthetic; Drug: Fluid administration; Procedure: Low-tidal volume ventilation

INTERVENTIONS:
Drug: Fluid resuscitation or amine administration — Fluid administration or amine administration if deemed necessary by the attending physician. Haemodynamics will be monitored through noninvasive cardiac output assessment by arterial pulse contour analysis
Drug: General anesthetic — Total intravenous anesthesia with a standard protocol
Drug: Fluid administration — 3-5 ml/kg of balanced crystalloids will be administered throughout the whole surgical procedure
Procedure: Low-tidal volume ventilation — Volume-control ventilation with tidal volume=7 ml/kg of predicted body weight for the entire surgical procedure. Respiratory rate will be set to maintain EtCO2 within a physiological range and kept unchanged for the entire duration of the study
Procedure: Scheduled recruiting maneuvers — Pressure-control ventilation inspiratory pressure=10 cmH2O. Steplike 5-cmH2O-PEEP increase every 30 seconds to achieve a peep of 35 cmH2O, followed by 5-cmH2O-PEEP reduction every 30 seconds to set PEEP
  Arms: PEEP12 + RM; PEEP2 + RM; PEEP7 + RM

SUMMARY:
Low-tidal volume ventilation is arising as a tool to optimize the ventilatory management and to improve clinical outcome in patients undergoing general anesthesia for abdominal surgery.

A recent large randomized controlled trial failed to detect a significant difference between two different approaches for ensuring adequate lung recruitment (PEEP=12 cmH2O + scheduled recruiting maneuvers vs. PEEP 2 cmH2O) during protective ventilation. Thus, in patients undergoing open abdominal surgery and receiving low-tidal volumes, the effects of different positive end-expiratory pressure (PEEP) levels and recruiting maneuvers remain to be established.

Design: prospective, cross-over, physiological trial.

PURPOSE To assess the physiological effects of different PEEP levels with or without scheduled recruiting maneuvers in patients undergoing general anesthesia for open abdominal surgery and receiving low-tidal volume ventilation.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II patients
* scheduled for open abdominal surgery (major gastrointestinal surgery: duodeno-cephalo-pancreatectomy, gastrectomy, hemi-colectomy; gynecological surgery; oncologic surgery)
* Expected duration of surgery >= 150 minutes

Exclusion Criteria:

* Pregnancy
* BMI>30 kg/m^2
* hepatic surgery
* Cardiac failure NYHA>2
* History of chronic respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Driving Pressure | At the end of each 40-minute step
  Respiratory system elastic pressure (Plateau pressure-total PEEP)

SECONDARY OUTCOMES:
Lung strain | At the end of each 40-minute step
  Lung static and dynamic strain
Dead space | At the end of each 40-minute step
  Approximated as the difference between End-tidal CO2 and PaCO2 divided by PaCO2
Oxygenation | At the end of each 40-minute step
  PaO2/FiO2
Lung recruitment | At the end of each 40-minute step
  % (lung recruitment/change in end-expiratory lung volume)
Lung overdistension due to PEEP | At the end of each 40-minute step
  % (lung overdistension/change in end-expiratory lung volume)
Functional residual capacity | At the end of each 40-minute step
  Change in functional residual capacity due to PEEP, measured with the Nitrogen washin-washout technique
Heart rate | At the end of each 40-minute step
  heart rate
Blood pressure | At the end of each 40-minute step
  Arterial blood pressure
Stroke volume | At the end of each 40-minute step
  Stroke volume, measured by pulse contour analysis
Stroke volume variation | At the end of each 40-minute step
  Stroke volume variation, measured by pulse contour analysis
Cardiac Output | At the end of each 40-minute step
  Stroke volume x heart rate
Fluid requirements | At the end of each 40-minute step
  Fluid bolus requirements, according to the decision of the attending physician blinded to the design of the study
Vasoactive agents | At the end of each 40-minute step
  Vasoactive agents requirements, according to the decision of the attending physician blinded to the design of the study
Adverse events | At the end of each 40-minute step
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- General surgery OR, A. Gemelli hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided